CLINICAL TRIAL: NCT07264127
Title: I-arch in Action: Early Clinical Impact From a Randomized Controlled Trial
Brief Title: Clinical Performance of the I-arch System During the Initial Stage of Orthodontic Treatment
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tabark H. Omran (Other)
Collaborators: University of Baghdad (Other)
Responsible Party: Sponsor-Investigator, Tabark H. Omran, Principal investigator, University of Baghdad
Organization: University of Baghdad (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ORTHO-UOB-2025
Record Dates: First submitted 2025-11-23; First posted 2025-12-04 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Effectiveness of I-arch System
Keywords: Archwire; Teeth alignment; Crowding; Orthodontics; Clinical trial; I-arch
MeSH Terms: conditions — Crowding

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: I-arch system (Experimental): Intervention: Use of 0.016×0.014-inch copper nickel titanium arch wire during the alignment stage.
  Interventions: Device: The use of 0.016×0.014 copper nickel titanium arch wire during the alignment stage.
- Arm 2: MBT arch wire system (Active Comparator): Intervention: Use of 0.014- then 0.016-inch heat-activated nickel titanium arch wire during the alignment stage.
  Interventions: Device: Use of 0.014- then 0.016-inch heat-activated nickel titanium arch wire during the alignment stage.

INTERVENTIONS:
Device: The use of 0.016×0.014 copper nickel titanium arch wire during the alignment stage. — Teeth alignment using an initial arch wire with a rectangular switched cross-section since the beginning of the treatment.
  Arms: Arm 1: I-arch system
Device: Use of 0.014- then 0.016-inch heat-activated nickel titanium arch wire during the alignment stage. — Teeth alignment using initial arch wires with round cross sections.
  Arms: Arm 2: MBT arch wire system

SUMMARY:
The goal of this clinical trial is to learn if the I-arch system works to align the moderately misaligned teeth in patients seeking orthodontic treatment. it aims to answer the following questions:

* Does I-arch system increase the rate of teeth alignment?
* Does I-arch system produce significant changes in arch width and incisors inclination?
* Does I-arch system decrease the intensity of patient-reported pain and root resorption? Researchers will compare the effectiveness of the I-arch and MBT arch wire system.

DETAILED DESCRIPTION:
This study will be a multicenter non-stratified prospective randomized clinical trial designed as a blinded, parallel group trial with equal randomization (1:1 allocation ratio). It will be conducted at multiple orthodontic centers. Initially, the eligibility of the patients to participate in this study will be evaluated by the investigator. Verbal information about the nature of study will be supplied for those who will satisfy the inclusion criteria to obtain their preliminary approval. Then the patient information sheet and consent form will be given to the patients to read carefully at home to decide whether they will participate in the study at the following visit. Patient assent/parental consent will be taken for participants below 18 years. If the patients have any queries regarding the study, the investigator should resolve it on the following visit.

Orthodontic treatment will be conducted using a straight wire appliance. MBT prescription brackets with 0.018-inch slot (Microfit™, SIA Orthodontic Manufacturer, Italy) will be used. With the aid of a height gauge, standardized bracket placement will be achieved. The technique will begin with a 10-second prophylactic procedure to clean and polish the teeth surfaces with pumice and a rubber cup using a slow-speed handpiece. Then, teeth will be rinsed with water and dried with oil-free air spray for 30 seconds. For the purpose of standardization, bonding procedure will be as followed:

* The enamel surface will be etched with 37% phosphoric acid gel for 30 seconds.
* The acid etchant will be rinsed off with water spray thoroughly.
* The tooth surface will be dried by air spray until the white frosty appearance of the etched surface is seen.
* A thin layer of Light Bond™ Sealant (Reliance®, Itasca, USA) will be applied on the etched enamel surface for one minute, then air will be applied for 5 seconds.
* Brackets and tubes will be bonded using Light Bond™ light cure orthodontic adhesive (Reliance®, Itasca, USA) which applied on their bases and light-cured above interproximal contacts at a distance of 2-3 mm (5 seconds mesially and 5 seconds distally for brackets and 10 seconds mesially and 10 seconds occlusally for molar tubes).

Arch wire sequence for each group will be as follows:

1. I-arch system group (I-arch™ Orthodontic System, SIA Orthodontic Manufacturer, Italy. (

   • 0.016×0.014-inch copper nickel titanium.
2. MBT arch wire system group (Thermal NiTi™, SIA Orthodontic Manufacturer, Italy)

   * 0.014-inch heat-activated nickel titanium.
   * 0.016-inch heat-activated nickel titanium. A standardized protocol will be followed during the treatment for all the participants. At the day of bonding, 0.016×0.014 copper nickel titanium arch wire will be placed for the I-arch group and religated every four weeks. While, for the MBT group, 0.014-inch heat-activated nickel titanium arch wire will be placed at the day of bonding, then after 8 weeks it will be replaced by the 0.016-inch heat-activated nickel titanium arch wire for another 8 weeks (both will be religated every four weeks). Elastomeric modules will be used for ligating the wire to the brackets. If any bracket debonding occurs throughout the course of the treatment, it should be bonded again during 24 hours. Otherwise, the participant will be excluded from the trial. Since this study will be performed during the initial phase of treatment, no deviation from the protocol of treatment will be accepted (such as adding additional arch wire in the sequence or using power chain). Digital scan for the maxillary and mandibular arches will be taken pre-treatment and after 4, 8, 12 and 16 weeks, and a digital model will be obtained which will be used to measure Little's irregularity index, the intercanine and intermolar widths. Lateral cephalometric radiograph and periapical radiographs (for the maxillary and mandibular central incisors) will be taken pre-treatment and after 16 weeks. Lateral cephalometric radiographs will be used to measure the inclination of the maxillary and mandibular incisors. While the periapical radiographs will be used to assess the root resorption of the maxillary and mandibular central incisors. The participants will be supplied with a visual analog scale (0-10) to record their pain perception during the first seven days following the first wire placement. At the end of the trial, the treatment will continue as prescribed.

ELIGIBILITY:
Inclusion Criteria:

1. Moderate crowding of mandibular anterior teeth (3-6 mm) according to Little's irregularity index (LII) in patients with age of 12 years or older.
2. Full complement of permanent dentition should be present, except for the third molars.
3. Brackets should be placed on maxillary and mandibular anterior teeth without any interference by the existing overbite and overjet.
4. The maxillary and mandibular incisors should not be previously subjected to trauma or root resorption.

Exclusion Criteria:

1. Patients with history of previous orthodontic treatment.
2. Severe maxillary and mandibular anterior crowding which is greater than 6 mm (LII).
3. Presence of teeth that are severely misaligned out of the dental arch and cannot be engaged with the aligning arch wire.
4. Prescence of periodontally compromised teeth and previous loss of attachment.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
The rate of alignment | 16 weeks
  Alignment rate will be measured using Little's Irregularity Index on digital dental models.

SECONDARY OUTCOMES:
The amount of inclination of the incisors | 16 weeks
  Maxillary and mandibular incisors inclination will be measured on lateral cephalometric radiographs.
The change in the width of dental arches | 16 weeks
  Maxillary and mandibular intermolar and intercanine widths will be measured on digital dental models.
The amount of root resorption | 16 weeks
  the root resorption of the maxillary and mandibular central incisors will be assessed on periapical radiographs using the long cone paralleling technique.
The intensity of pain | Throughout the seven days following the insertion of the first arch wire
  Pain intensity will be measured using visual analog scale.

CONTACTS AND LOCATIONS:
Overall Officials: Yassir Yassir, PhD, Study Director — College of dentistry/ Baghdad university

IPD SHARING:
Plan to Share IPD: No
For the purpose of maintaining the confidentiality of the participants and the associated restrictions imposed by the ethics committee, we choose not to share IPD. However, IPD can be shared with journal editor upon request during the study publication.